CLINICAL TRIAL: NCT06094816
Title: Forebrain Electroneutral Transporters in Salt-sensitive Hypertension: an MRI Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2053776; R01HL163906 (NIH)
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Salt-Sensitivity of Blood Pressure
MeSH Terms: interventions — Furosemide; Diuretics

STUDY DESIGN:
Intervention Model Description: Double blind randomized cross-over
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salt Resistant Adults (Experimental): Adults who experience minimal BP change during dietary sodium challenge
  Interventions: Drug: Furosemide (Diuretic); Other: Hypertonic Saline Infusion
- Salt Sensitive (Experimental): Adults who experience increased BP (mean arterial pressures >5mmHg) during dietary sodium challenge
  Interventions: Drug: Furosemide (Diuretic); Other: Hypertonic Saline Infusion

INTERVENTIONS:
Drug: Furosemide (Diuretic) — The diuretic furosemide will be given during a 3% hypertonic saline infusion to examine blockade of the NKCC2.
  Other Names: Lasix
Other: Hypertonic Saline Infusion — 3% Hypertonic saline infusion to acutely increase sodium and osmolality

SUMMARY:
The overall objective of this project is to identify the key salt-sensing regions of the brain and determine the underlying mechanism of sodium sensing. The investigators will assess how the brain responds to an acute increase of salt in the blood using MRI. This will be done during a 30-minute infusion of a saline solution containing 3% salt. One trial will be conducted with a salt sensing channel blocker and one trial without the salt sensing channel blocker. This will help to assess the role of a specific salt sensing channel in the brain. Salt sensitivity of BP will be assessed using 7-day dietary feeding where participants will be given food to consume for 7-days. Comparisons will be made between salt resistant (no change in blood pressure going from low to high salt diets) and salt sensitive adults (a change in blood pressure going from low to high salt diets). The investigators think the changes in MRI will be greater in salt sensitive compared to salt resistant subjects.

DETAILED DESCRIPTION:
The ability of the brain to sense changing sodium levels in the blood is critical in mediating the neurohumoral responses to hypernatremia, however, the mechanisms underlying sodium sensing in humans is poorly understood. The purpose of this study is to identify key sodium-sensing regions of the human brain in middle-aged men and women with high blood pressure and determine if the Na-K-2Cl co-transporter (NKCC2) mediates the neurohumoral response to acute hypernatremia. The investigators plan on comparing these central sodium responses to acute hypernatremia between salt-sensitive and salt-resistant adults. In this randomized double-blinded crossover study subjects will have a 3% NaCl (hypertonic saline) infusion with or without NKCC2 antagonism (furosemide). Completion of this project will increase the understanding of blood pressure regulation, which has major public health implications.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 40 years or < 60 years
* Blood pressure: > 100/60 mmHg or < 140/90 mmHg
* BMI: > 18.5 kg/m2 or < 30 kg/m2
* Serum potassium: > 3.5 mmol/L or < 5.5 mmol/L
* No history of cardiovascular, renal, metabolic, or neurological disease

Exclusion Criteria:

* Age: < 40 years or > 60 years
* Blood pressure: < 100/60 mmHg or > 140/90 mmHg
* BMI: < 18.5 kg/m2 or > 30 kg/m2
* Serum potassium: < 3.5 mmol/L or > 5.5 mmol/L
* Abnormal ECG
* History of - cardiovascular, cancer, metabolic, respiratory, renal disease
* Hormone replacement therapy
* Current tobacco or nicotine use
* Pregnant or nursing mothers
* Major brain injury (concussions do not count)
* Clinically diagnosed psychiatric or neurological disorder
* Clinically diagnosed anxiety or depression
* Psychiatric, neurological, anxiety or depression medications
* Hypertension medications
* Sulfonamide drug allergy
* Contra-indications to MRI (implants, metal, etc)
* Claustrophobia

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Bold fMRI | 1 hour
  Intensity of sodium sensing regions of the brain

SECONDARY OUTCOMES:
Blood Pressure | 1 hour
  Systolic and Diastolic Blood pressure responses to hypertonic saline

OTHER OUTCOMES:
Sympathetic Nerve Activity | 1 hour
  sympathetic bursts per minute

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No